CLINICAL TRIAL: NCT05506436
Title: Evaluation of an Implementation Strategy of mHealth Intervention for the Promotion of Healthy Lifestyles in Primary Healthcare (E-VIDAPP Pilot Study)
Brief Title: Evaluation of an Implementation Strategy of mHealth Intervention to Promote Healthy Lifestyles (E-VIDAPP Pilot Study)
Acronym: E-VIDAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IBYE2100001
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-08

CONDITIONS: Healthy Lifestyle; Nursing
Keywords: Implementation science; Health Promotion; Primary Health Care; mHealth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation group (Experimental): Four sessions are conducted with the nurses of the center assigned to the intervention group to agree on the implementation strategy together with the professionals. Once the strategy is defined, the implementation of the intervention will be launched in this group for 6 months. After this period, the final evaluation will be carried out, as well as a qualitative evaluation through a focus group.
  Interventions: Device: Evident 3; Other: Implementation strategy
- Control group (Active Comparator): A single session will be scheduled to introduce the nurses of the center assigned to this group to the EVIDENT 3 intervention, and access and downloading will be allowed for free use in their practice.
  Interventions: Device: Evident 3

INTERVENTIONS:
Device: Evident 3 — It consists of brief 5-minute counselling on general physical activity recommendations and explaining the plate method for a balanced diet. Also, it includes the Evident 3 application, which is a daily dietary log that provides information on calories and diet composition and shows a reminder of the 10000 steps/day.
Other: Implementation strategy — Four sessions have been designed to obtain the implementation strategy:
  First session: Presentation of the Evident 3 application and its results in clinical trials. Training in the use of the application and identification of possible areas for improvement.
  Second session: Presentation of evidence-based practices on the management of obesity in Primary Care. Consensus selection of those related to health promotion and mHealth. Sharing of possible lines of improvement of the care offered in the practice.
  Third session (optional): Intervention on those components (coherence, cognitive participation, collective action and reflective follow-up) of the NOMAD questionnaire, if very low scores are obtained.
  Fourth session: Brainstorming on possible strategies for the implementation of the Evident 3 intervention. Analysis and evaluation of these strategies and determination of a common strategy for their implementation.
  Arms: Implementation group

SUMMARY:
The translation of beneficial interventions for the population into professional practice represents a constant challenge. Moreover, implementation of this evidence into clinical practice has been limited to date. Therefore, the aim of this pilot study is to identify the critical factors and barriers that may influence the implementation of a digital intervention for the promotion of exercise and a healthy diet in primary care and its implementation through a pilot study with a strategy agreed with nursing professionals in a health centre.

DETAILED DESCRIPTION:
DESIGN: Pilot study with mixed methodology (quantitative and qualitative). A pre-implementation visit was performed to evaluate the variables of the study. After completion of this visit, intervention and control groups are randomly assigned. Training and participatory sessions are carried out in the intervention group. After these sessions, the EVIDENT 3 intervention is implemented for 6 months in the nursing offices. After this 6-month period, the final evaluation will be carried out, as well as a focus group in the intervention group.

STUDY POPULATION: The study participants are the nursing professionals working in the health centers that have been working in one of the selected centers for at least 6 months prior to the start of the study, with permanence in the same until the end of the study, who agree to participate and who sign the informed consent form.

IMPLEMENTATION STRATEGY

1. Specific intervention in the intervention group: 4 training sessions on the following topics: 1-Evident intervention, 2-Evidence-based clinical practice, 3- Main components of Normalization Process Theory, 4- Implementation strategies.
2. Intervention to be implemented: The intervention to be explained to the professionals is the EVIDENT 3 intervention, which proves its efficacy previously. It consists of brief advice on nutrition, using the plate method (50), and advice on physical activity based on the current recommendations of at least 30 minutes of moderate activity 5 days a week, or 20 minutes of vigorous activity, 3 days a week. In addition, the EVIDENT 3 mobile app is included, which was designed to allow self-reporting of daily nutrition. Once the user enters all the information, the app integrates all the data to create personalized recommendations and weight loss goals.
3. Qualitative research: In the final evaluation of the study, a focus group discussion will be conducted from a phenomenological perspective, only with participants from the intervention group. The sampling will be theoretical in order to achieve maximum discursive plurality. A random selection of the participants who have marked the option to participate in the qualitative study in the consent form will be contacted.

STRUCTURE OF THE STUDY VISITS:

Pre-implementation visit: Inclusion criteria, explanation of the project, informed consent and baseline assessment of the study variables.

Assignment of study groups (intervention and control). Implementation: 4 training sessions in the intervention group . After these sessions, the implementation will be piloted in real conditions for a 6-months period.

Final visit: Post-implementation evaluation will be done at the end of the implementation (6 months) to evaluate changes in the study variables in both groups. A discussion group will be held in the intervention group to evaluate the experience of the implementation

ELIGIBILITY:
Inclusion Criteria:

* Nurses who have been working in one of the selected centers for at least 6 months prior to the start of the study, with permanence until the end of the study.
* Acceptance to participate and sign the informed consent form

Exclusion Criteria:

* Nurses who have been working at the center for less than 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Use of the intervention EVIDENT 3 | 6 months
  It will be evaluated by the number of downloads of the application from the platform created for this purpose in RedCap per primary health centre.
Number of obesity-related activities in primary health care | 6 months
  It will be evaluated with the clinical practice questionnaire in the management of obesity, which evaluates the frequency (weekly, monthly or never) of 7 activities that are performed in the office related to obesity. This questionnaire has no cut-off point.

SECONDARY OUTCOMES:
Level of nurses' self-efficacy in obesity management | 6 months
  It will be evaluated by the Self-efficacy in obesity management Questionnaire, with 23 items on a Likert scale with 4 possible answers. This questionnaire has no cut-off point.
Level of acceptance of the implementation of the intervention | 6 months
  Measured with the Normalisation Measure Development questionnaire (NoMAD), which evaluates the implementation of complex health interventions. It consists of 23 questions grouped into four constructs: C1 Coherence (4 questions); C2 Cognitive involvement (4 questions); C3 Collective action (7 questions); C4 Reflective monitoring or "Evaluation"(5 questions) and 3 standardization questions.This questionnaire has no cut-off point.
Level of the willingness of healthcare organizations to change clinical practice | 6 months
  It will be evaluated with the Organizational Readiness for Knowledge Translation (OR4KT) questionnaire. It assesses 6 domains (organizational climate for change, contextual and organizational factors, change content, leadership, organizational support and motivation) through 59 items with a 5-choice Likert scale. A score greater than 64 indicates a greater willingness to change clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Research Unit of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided